CLINICAL TRIAL: NCT03928912
Title: Risk Factors for Post-Operative Nonunion of Tibial Shaft Fractures Based on a Path Analysis Model: A Case-Control Study
Brief Title: Risk Factors for Post-Operative Nonunion of Tibial Shaft Fractures Based on a Path Analysis Model
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: I2019001035
Record Dates: First submitted 2019-04-21; First posted 2019-04-26 (Actual); Last update posted 2019-04-26 (Actual); Status verified 2019-04

CONDITIONS: Nonunion of Fracture of Tibia (Diagnosis)
Keywords: nonunion; tibial shaft fracture; path analysis model
MeSH Terms: conditions — Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- without fracture nonunion: The patients who undergone surgery after tibial shaft fracture did not exist fracture nonunion
- with fracture nonunion: The patients who undergone surgery after tibial shaft fracture existed fracture nonunion

SUMMARY:
Tibial shaft fractures is common long tubular fracture that account for about 13.7% of all fractures. And the incidence of nonunion of tibial shaft fracture varied from 1% to 80%. This study aimed to confirm the risk factors of nonunion of tibial shaft fracture. Moreover, the investigators hope to establish the clinical pathway of various risk factors for fracture nonunion and affirm the importance of different risk factors.

DETAILED DESCRIPTION:
Tibial shaft fractures is common long tubular fracture that account for about 13.7% of all fractures. And the incidence of nonunion of tibial shaft fracture varied from 1% to 80%. The investigators retrospectively analyzed the demographics of these participants in our hospital that occur long tubular fracture. One group is participants that existed fracture nonunion. And the other group is the participants that did not exist fracture nonunion. The investigators recorded twelve variables and confirm the risk factors by uni-variate Logistic regression analysis. Moreover, the investigators hope to establish the clinical pathway of various risk factors for fracture nonunion and affirm the importance of different risk factors.

ELIGIBILITY:
Inclusion Criteria:

* The tibial shaft fracture was caused by trauma.

Exclusion Criteria:

* The tibial shaft fracture was caused by tumor, infection and other reasons.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The population came from The Second Affiliated Hospital of Zhejiang University.
Sampling Method: Probability Sample
Enrollment: 234 (Actual)
Dates: Start 2019-02-02 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-10 (Actual)

PRIMARY OUTCOMES:
the Gustilo type of the open fracture | the outcome of the Gustilo type can acquire within 1 week.
  the Gustilo type of the open fracture can be divided into three types. And the type I is the open fractures with wounds that is clean and smaller than 1cm. Type II is the the open fractures with wounds that is moderately unclean and bigger than 1cm, which also has a wide soft tissue injury. Type III is the all open fractures that accompany with severe soft tissue injury and pollution.

CONTACTS AND LOCATIONS:
Overall Officials: Jian'an Wang, Ph.D, Study Chair — Zhejiang University
Locations (1):
- Institutional Review Board of The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China